CLINICAL TRIAL: NCT06037447
Title: A Prospective Controlled Study for the Treatment Effect of Different Intervention Strategies for Pediatric Mitral Regurgitation--A Multicenter Prospective Cohort Study of Innovative Strategies for Mitral Valve Repair
Brief Title: Study of Innovative Strategies for Mitral Valve Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Shanghai Children's Medical Center (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Guangzhou Women and Children's Medical Center (Other); Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Shoujun Li, Director of Congenital Heart Surgery Center, China National Center for Cardiovascular Diseases
Other Study IDs: 2022-GSP-GG-19-2
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Congenital Mitral Insufficiency
Keywords: congenital heart disease; mitral regurgitation; mitral valve repair
MeSH Terms: conditions — Heart Defects, Congenital; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standardized Group: Patients in this group will undergo standardized strategy during mitral repair surgeries, including subvalvular apparatus rehabilitation, leaflets repair and annuloplasty.
  Interventions: Procedure: 3-steps standardized repair-oriented strategy
- Annuloplasty Group: Patients in this group will undergo annuloplasty only during mitral repair surgeries.

INTERVENTIONS:
Procedure: 3-steps standardized repair-oriented strategy — 3-steps standardized repair-oriented strategy, including subvalvular apparatus rehabilitation (leaflet plication if chordae absent on leaflet margin, mal-connected chordae resection if chordae mal-connected to leaflet body, papillary muscle splitting if short chordae or dysplastic or fused papillary muscle etc.), leaflets repair (leaflets plication if functional leaflet prolapse, leaflet cleft closure and patch augmentation for anatomical leaflet defect, etc.) and annuloplasty (posterior annuloplasty for annular dilatation and shallow leaflet coaptation, etc.)
  Groups: Standardized Group

SUMMARY:
The goal of this observational study is to compare the safety and effectiveness of a 3-steps standardized repair-oriented strategy with annuloplasty only in pediatric patients with mild to moderate mitral valve regurgitation.

The main questions it aims to answer are:

* Can 3-steps standardized repair-oriented strategy improve both left ventricular and mitral valve function in pediatric patients with mild to moderate mitral valve regurgitation?
* Can surgical complications caused by the 3-steps standardized repair-oriented strategy be non-inferior (clinically acceptable) to annuloplasty only? Participants will be assigned to either the Standardized Group (including subvalvular apparatus rehabilitation (leaflet plication if chordae absent on leaflet margin, mal-connected chordae resection if chordae mal-connected to leaflet body, papillary muscle splitting if short chordae or dysplastic or fused papillary muscle etc.), leaflets repair (leaflets plication if functional leaflet prolapse, leaflet cleft closure and patch augmentation for anatomical leaflet defect, etc.) and annuloplasty (posterior annuloplasty for annular dilatation and shallow leaflet coaptation, etc.)) or the Annuloplasty Group (annuloplasty only during mitral repair surgeries. Additionally, echocardiography, electrocardiograms, and measurements of N-terminal pro-brain natriuretic peptide (NT-proBNP) were conducted before the initiation of surgery and at 1 months, 3 months, and 6 months after mitral repair.

Researchers will compare the Standardized Group and the Annuloplasty Group to see if the recurrence rate of moderate to severe mitral valve regurgitation, as assessed by echocardiography after 6 months of surgery, is lower in the former than in the latter.

ELIGIBILITY:
Inclusion Criteria:

* < 14 years old
* had not undertake mitral valve surgery before
* moderate to severe mitral regurgitation

Exclusion Criteria:

* moderate to severe mitral regurgitation which concommitant with other cardiac malformation which can not be correct or can only perform palliative surgery
* concommitant with mitral stenosis
* ischemic mitral regurgitation (for example, concommitant with anomalous origin of coronary artery)
* Barlow syndrome
* dysplasia of mitral leaflet
* complete/Partial endocardial cushion defect
* common atrioventricular valve
* atrioventricular common channel
* cardiomyopathy
* other mitral valve surgery contraindications

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under the age of 14 with moderate to severe mitral valve regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-05 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the recurrence rate of moderate to severe mitral valve regurgitation | after 6 months of surgery
  During follow-up visits, echocardiographic examination is conducted to measure the degree of mitral valve regurgitation. If it falls within the moderate to severe range, it is recorded as a recurrence.

SECONDARY OUTCOMES:
Improvement in symptoms | after 6 months of surgery
  Based on patient and caregiver descriptions, if symptoms such as chest discomfort, shortness of breath, and delayed development show improvement following physical activity, it is recorded as an improvement in symptoms.
Change in left ventricular function | after 6 months of surgery
  Based on the echocardiogram, measurements are taken for left ventricular ejection fraction.
Change in left ventricular function | after 6 months of surgery
  Based on the echocardiogram, measurements are taken for left ventricular end-diastolic diameter.
NT-proBNP level | after 6 months of surgery
  The trend in NT-proBNP levels.
Incidence rate of surgical complications | after 6 months of surgery
  Incidence rate of surgical complications, including infection, low cardiac output, arrhythmia, cardiac insufficiency, delayed sternal closure, thromboembolism and bleeding events, neurological complications(stroke, seizures and intracerebral hemorrhage).

CONTACTS AND LOCATIONS:
Overall Officials: Shoujun Li, MD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No